CLINICAL TRIAL: NCT06291428
Title: Raman Spectroscopy Compared to Flow Cytometry as a Method for Assessing Measurable Residual Disease in Patients With Acute Lymphoblastic Leukemia
Brief Title: Raman Spectroscopy Compared to Flow Cytometry
Status: Recruiting | Type: Observational
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Lauro Fabian Amador Medina, Dr., Hospital Regional de Alta Especialidad del Bajio
Other Study IDs: F-CNIC-2024-007
Record Dates: First submitted 2024-02-23; First posted 2024-03-04 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Raman spectroscopy: Patients with acute lymphoblastic leukemia, in assessment for measure residual disease.
  Interventions: Diagnostic Test: Raman spectroscopy
- flow citometry: Patients with acute lymphoblastic leukemia, in assessment for measure residual disease.
  Interventions: Diagnostic Test: Raman spectroscopy

INTERVENTIONS:
Diagnostic Test: Raman spectroscopy — Raman spectroscopy is proposed as a potential technique for MRD measurement, which is based on the inelastic scattering of light that occurs when it interacts with matter, causing optical scattering, where a portion of the radiation changes its wavelength (by Raman effect). By analyzing the inelastically scattered light, we can obtain a Raman spectrum formed by the intensity of the scattered light as a function of its vibration frequency, thus obtaining information about the biochemical composition of a biological sample.

SUMMARY:
The detection of MRD is associated with an increased risk of relapse and adverse prognosis in all patient groups diagnosed with acute lymphoblastic leukemia (ALL). However, it has a sensitivity level that detects one leukemic cell in 10,000 normal cells, along with other disadvantages such as the need for a panel of fluorescent antibodies for MRD detection, and its measurement is not standardized in many centers. New determination techniques may be necessary for MRD evaluation. Raman spectroscopy is proposed as a potential technique for MRD measurement, which is based on the inelastic scattering of light that occurs when it interacts with matter, causing optical scattering, where a portion of the radiation changes its wavelength (by Raman effect).

Objectives:

MAIN OBJECTIVE:

To evaluate the presence of MRD in patients with ALL by comparing a standard evaluation method using flow cytometry with a new proposed method using Raman spectroscopy.

SPECIFIC OBJECTIVES:

* To assess the presence of MRD using flow cytometry in patients with ALL.
* To assess the presence of MRD using Raman spectroscopy in patients with ALL.
* To perform a comparison between the MRD measurement techniques by determining sensitivity, specificity, positive predictive value, and negative predictive value.
* To establish the validation of using Raman spectroscopy as a method for MRD evaluation.

Study Design:

An observational, cross-sectional, comparative, and diagnostic test study will be conducted on bone marrow aspirate samples from adult and pediatric ALL patients to evaluate the presence of MRD using Raman spectroscopy, comparing the results of this technique with those obtained using flow cytometry. As a diagnostic test study, sensitivity, specificity, positive predictive value, and negative predictive value will be evaluated. The study will be conducted on adult and pediatric patients diagnosed with acute lymphoblastic leukemia treated at the hemato-oncology department of the UMAE No. 1 National Medical Center Bajio and the UMAE Hospital Gynecology-Pediatrics No. 48.

Inclusion Criteria:

Patients diagnosed with ALL for whom MRD determination is clinically necessary will be included in the study. Their results will be evaluated using the gold standard, flow cytometry, and compared with results obtained through Raman spectroscopy.

DETAILED DESCRIPTION:
The assessment of measurable residual disease (MRD) is a frequent practice in the management of acute lymphoblastic leukemia (ALL). The detection of MRD is associated with an increased risk of relapse and adverse prognosis in all patient groups diagnosed with ALL. The three approved methods for MRD measurement are flow cytometry, polymerase chain reaction (PCR) of specific mutations, and next-generation sequencing (NGS). Of these, flow cytometry is the most used method in clinical practice. However, it has a sensitivity level that detects one leukemic cell in 10,000 normal cells, along with other disadvantages such as the need for a panel of fluorescent antibodies for MRD detection, and its measurement is not standardized in many centers. New determination techniques may be necessary for MRD evaluation. Raman spectroscopy is proposed as a potential technique for MRD measurement, which is based on the inelastic scattering of light that occurs when it interacts with matter, causing optical scattering, where a portion of the radiation changes its wavelength (by Raman effect). By analyzing the inelastically scattered light, we can obtain a Raman spectrum formed by the intensity of the scattered light as a function of its vibration frequency, thus obtaining information about the biochemical composition of a biological sample.

Objectives:

MAIN OBJECTIVE:

To evaluate the presence of MRD in patients with ALL by comparing a standard evaluation method using flow cytometry with a new proposed method using Raman spectroscopy.

SPECIFIC OBJECTIVES:

* To assess the presence of MRD using flow cytometry in patients with ALL.
* To assess the presence of MRD using Raman spectroscopy in patients with ALL.
* To perform a comparison between the MRD measurement techniques by determining sensitivity, specificity, positive predictive value, and negative predictive value.
* To establish the validation of using Raman spectroscopy as a method for MRD evaluation.

Study Design:

An observational, cross-sectional, comparative, and diagnostic test study will be conducted on bone marrow aspirate samples from adult and pediatric ALL patients to evaluate the presence of MRD using Raman spectroscopy, comparing the results of this technique with those obtained using flow cytometry. As a diagnostic test study, sensitivity, specificity, positive predictive value, and negative predictive value will be evaluated. The study will be conducted on adult and pediatric patients diagnosed with acute lymphoblastic leukemia treated at the hemato-oncology department of the UMAE No. 1 National Medical Center Bajio and the UMAE Hospital Gynecology-Pediatrics No. 48.

Inclusion Criteria:

Patients diagnosed with ALL for whom MRD determination is clinically necessary will be included in the study. Their results will be evaluated using the gold standard, flow cytometry, and compared with results obtained through Raman spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ALL for whom MRD determination is clinically necessary will be included in the study.

Exclusion Criteria:

* Patients without ALL

Ages: 2 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
measurable residual disease | up to 1 year
  To evaluate the presence of MRD in patients with ALL by comparing a standard evaluation method using flow cytometry with a new proposed method using Raman spectroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional Alta Especialidad Bajio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided